CLINICAL TRIAL: NCT03811288
Title: A Non-interventional Cross-sectional Study to Capture the Prevalence of Cardiovascular Disease in Patients With Type 2 Diabetes - an International Observation
Brief Title: An International Survey of the Occurrence of Cardiovascular Disease Among Patients With Type 2 Diabetes
Acronym: CAPTURE-IO
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4446; U1111-1215-4005 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-01-18; First posted 2019-01-22 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with type 2 diabetes mellitus (T2DM): T2DM patients being managed in both primary and specialist care in 10 selected countries.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No specific intervention is studied. All anti-diabetic and CV medication will be prescribed at the physician's discretion under routine clinical practice conditions.

SUMMARY:
The purpose of the study is to register the occurrence of cardiovascular disease among type 2 diabetes patients across ten countries across the world. Participants will be asked to give information about their health. Participants will continue their normal way of life and will not get any medication other than prescribed to them by their doctor. Participants' participation will be one day/one visit at their doctor. The study will last for about 6 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedures related to recording of data according to protocol)
* Male or female, age more than or equal to 18 years at the time of signing informed consent (in Algeria more than or equal to 19 years; in Japan more than or equal to 20 years).
* Diagnosed with T2DM more than or equal to 180 days prior to the day of signing the informed consent

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Diagnosed with Type 1 diabetes
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients with known congenital heart disease/malformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male and female adults diagnosed with T2DM.
Sampling Method: Non-Probability Sample
Enrollment: 7548 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Participants with a history of established cardiovascular disease (CVD) | Day 1
  Participants having a history of established CVD, i.e. who have been diagnosed with any one of the following listed conditions (yes/no): Cerebrovascular disease, cardiovascular disease, symptomatic heart failure, asymptomatic heart failure, hospitalisation for heart failure, cardiac arrhythmia, aortic disease, peripheral artery disease or carotid artery disease.

SECONDARY OUTCOMES:
Participants with high risk of CVD according to the risk engine from the United Kingdom Prospective Diabetes Study (UKPDS) | Day 1
  Percentage of participants (yes/no). High risk: more than 20 percent over 10 years.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (135):
- Algeria (5):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Batna City
  - Novo Nordisk Investigational Site, Constantine
  - Novo Nordisk Investigational Site, Tiaret
  - Novo Nordisk Investigational Site, Tizi Ouzou
- Argentina (9):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Chacabuco
  - Novo Nordisk Investigational Site, Coronel Suárez
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Godoy Cruz
  - Novo Nordisk Investigational Site, Lanús Este
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Morón
- Australia (18):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, Brookvale, New South Wales
  - Novo Nordisk Investigational Site, Campbelltown, New South Wales
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
  - Novo Nordisk Investigational Site, Maroubra, New South Wales
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, Herston, Queensland
  - Novo Nordisk Investigational Site, Morayfield, Queensland
  - Novo Nordisk Investigational Site, North Ipswich, Queensland
  - Novo Nordisk Investigational Site, Sherwood, Queensland
  - Novo Nordisk Investigational Site, Victoria Point, Queensland
  - Novo Nordisk Investigational Site, Forest Hill, Victoria
  - Novo Nordisk Investigational Site, Moonee Ponds, Victoria
  - Novo Nordisk Investigational Site, Parkville, Victoria
  - Novo Nordisk Investigational Site, Preston, Victoria
  - Novo Nordisk Investigational Site, Ringwood, Victoria
  - Novo Nordisk Investigational Site, Fremantle, Western Australia
  - Novo Nordisk Investigational Site, Geelong
- Brazil (17):
  - Novo Nordisk Investigational Site, Fortaleza, Ceará
  - Novo Nordisk Investigational Site, Aparecida de Goiânia, Goiás
  - Novo Nordisk Investigational Site, Goiânia, Goiás
  - Novo Nordisk Investigational Site, Belo Horizonte, Minas Gerais
  - Novo Nordisk Investigational Site, Uberaba, Minas Gerais
  - Novo Nordisk Investigational Site, Campina Grande do Sul, Paraná
  - Novo Nordisk Investigational Site, Curitiba, Paraná
  - Novo Nordisk Investigational Site, Maringá, Paraná
  - Novo Nordisk Investigational Site, Passo Fundo, Rio Grande do Sul
  - Novo Nordisk Investigational Site, Porto Alegre, Rio Grande do Sul
  - Novo Nordisk Investigational Site, Campinas, São Paulo
  - Novo Nordisk Investigational Site, Santo André, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Tatuí, São Paulo
  - Novo Nordisk Investigational Site, Votuporanga, São Paulo
  - Novo Nordisk Investigational Site, Fortaleza
  - Novo Nordisk Investigational Site, São Paulo
- China (10):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Lanzhou, Gansu
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Guiyang, Guizhou
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Luzhou, Sichuan
  - Novo Nordisk Investigational Site, Nanchong, Sichuan
  - Novo Nordisk Investigational Site, Ningbo, Zhejiang
  - Novo Nordisk Investigational Site, Nanjing
- Israel (14):
  - Novo Nordisk Investigational Site, Bat Yam
  - Novo Nordisk Investigational Site, Beer-Sheva HaDarom
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Bnei Brak
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kiryat Bialik
  - Novo Nordisk Investigational Site, Nahariya
  - Novo Nordisk Investigational Site, Nazareth
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Raanana
  - Novo Nordisk Investigational Site, Safed
  - Novo Nordisk Investigational Site, Tel Aviv
- Japan (19):
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Ebina-shi, Kanagawa
  - Novo Nordisk Investigational Site, Fukushima
  - Novo Nordisk Investigational Site, Hamamatsu-Shi Shizuoka
  - Novo Nordisk Investigational Site, Hokkaido
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kawagoe-shi, Saitama
  - Novo Nordisk Investigational Site, Koshigaya-shi,Saitama
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Nishi-ku Sapporo
  - Novo Nordisk Investigational Site, Okawa-shi, Fukuoka
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Oyama-shi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Shimotsuke-shi, Tochigi
  - Novo Nordisk Investigational Site, Shinjyuku-ku Tokyo
- Mexico (26):
  - Novo Nordisk Investigational Site, Tijuana, Baja California Norte
  - Novo Nordisk Investigational Site, Monclova, Coahuila
  - Novo Nordisk Investigational Site, Celaya, Guanajuato
  - Novo Nordisk Investigational Site, León, Guanajuato
  - Novo Nordisk Investigational Site, Acapulco de Juárez, Guerrero
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Puerto Vallarta, Jalisco
  - Novo Nordisk Investigational Site, Zapopan, Jalisco
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Benito Juárez, México, D.F.
  - Novo Nordisk Investigational Site, Cuauhtémoc, México, D.F.
  - Novo Nordisk Investigational Site, Gustavo A. Madero, México, D.F.
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, San Luis Potosí City, San Luis Potosí
  - Novo Nordisk Investigational Site, Culiacán, Sinaloa
  - Novo Nordisk Investigational Site, Hermosillo, Sonora
  - Novo Nordisk Investigational Site, México, State of Mexico
  - Novo Nordisk Investigational Site, Ciudad Madero, Tamaulipas
  - Novo Nordisk Investigational Site, Aguascalientes
  - Novo Nordisk Investigational Site, Guadalajara
  - Novo Nordisk Investigational Site, Mexico City
  - Novo Nordisk Investigational Site, Monterrey
  - Novo Nordisk Investigational Site, Querétaro
  - Novo Nordisk Investigational Site, San Luis Potosí City
  - Novo Nordisk Investigational Site, Veracruz
- Saudi Arabia (5):
  - Novo Nordisk Investigational Site, Al Ihsa
  - Novo Nordisk Investigational Site, Buraidah
  - Novo Nordisk Investigational Site, Jeddah
  - Novo Nordisk Investigational Site, Riyadh
  - Novo Nordisk Investigational Site, Ta'if
- Turkey (Türkiye) (12):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Edirne
  - Novo Nordisk Investigational Site, Elâzığ
  - Novo Nordisk Investigational Site, Eskişehir
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Kayseri
  - Novo Nordisk Investigational Site, Malatya
  - Novo Nordisk Investigational Site, Tekirdağ
  - Novo Nordisk Investigational Site, Zonguldak

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://www.novonordisk-trials.com

REFERENCES:
- [Derived] Vencio S, Vianna AGD, da Silva MACF, Precoma DB. Contemporary (2019) prevalence of cardiovascular disease in adults with type 2 diabetes in Brazil: the cross-sectional CAPTURE study. Diabetol Metab Syndr. 2022 Jan 10;14(1):5. doi: 10.1186/s13098-021-00775-9. PMID 35012646
- [Derived] Mosenzon O, Alguwaihes A, Leon JLA, Bayram F, Darmon P, Davis TME, Dieuzeide G, Eriksen KT, Hong T, Kaltoft MS, Lengyel C, Rhee NA, Russo GT, Shirabe S, Urbancova K, Vencio S; CAPTURE Study Investigators. CAPTURE: a multinational, cross-sectional study of cardiovascular disease prevalence in adults with type 2 diabetes across 13 countries. Cardiovasc Diabetol. 2021 Jul 27;20(1):154. doi: 10.1186/s12933-021-01344-0. PMID 34315481